CLINICAL TRIAL: NCT00915486
Title: A Randomized, Multi-center, Controlled, Parallel Group, Dose Finding Study of the Efficacy and Safety of Topically Applied I-020201 as an Adjunct to Good Standard-of-care Versus Good Standard-of-care Alone in Patients With Chronic Diabetic Foot Ulcers
Brief Title: A Dose Finding Study of Topically Applied I-020201 as an Adjunct to Good Standard-of-care in Patients With Chronic Diabetic Foot Ulcers
Acronym: DFU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS I-020201/01
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic; ulcer; topical; PDGF; GSoC
MeSH Terms: conditions — Diabetic Foot; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Good Standard of Care (GSoC) (Experimental): Twice per week
  Interventions: Procedure: Good Standard of Care (GSoC)
- GSoC + vehicle (Experimental): Twice per week
  Interventions: Procedure: Good Standard of Care (GSoC); Biological: Vehicle
- GSoC + I-020201 (33microg) (Experimental): Twice per week
  Interventions: Procedure: Good Standard of Care (GSoC); Biological: I-020201
- GSoC + I-020201 (100microg) (Experimental): Twice per week
  Interventions: Procedure: Good Standard of Care (GSoC); Biological: I-020201
- GSoC + I-020201 (300microg) (Experimental): Twice per week
  Interventions: Procedure: Good Standard of Care (GSoC); Biological: I-020201

INTERVENTIONS:
Procedure: Good Standard of Care (GSoC) — Procedural treatment twice per week
Biological: Vehicle — Topical fibrin as an adjunct to GSoC twice per week
  Arms: GSoC + vehicle
Biological: I-020201 — Topical treatment with 3 different concentrations as an adjunct to GSoC twice per week
  Arms: GSoC + I-020201 (100microg); GSoC + I-020201 (300microg); GSoC + I-020201 (33microg)

SUMMARY:
Although major improvements in the management and treatment of diabetic foot ulcers have been made, the clinical and financial burden of such long-term wounds is still high and is likely to increase as the general population ages. The large population affected by diabetic foot ulcers and the high rates of failure ending with amputation even with the best therapeutic regimens have resulted in the development of new therapies. I-020201 is a bioactive therapy intended for topical treatment of hard-to-heal diabetic foot ulcers, stimulating the granulation tissue formation. This study aims to evaluate the safety and efficacy of I-020201 in adjunct to good standard of care in patients with chronic diabetic foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged ≥ 18 years
* given written informed consent
* female of childbearing potential with a negative result from the pregnancy test at screening who agrees to use an acceptable birth control method (hormonal or IUD) or abstinence throughout the trial
* Type 1 or Type 2 Diabetes mellitus with HbA1c =< 12%
* with only one diabetic foot ulcer on the foot to be treated on or below the ankle

Exclusion Criteria:

* pregnant or breast-feeding
* known or suspected allergies to any of the components of the I-020201
* uncontrolled anemia (Hb < 9 g/dL in females and < 10 g/dL in males)
* hypoalbuminemia (albumin < 3 g/dL)
* overtly infected target ulcer (as judged by investigator)
* highly exuding wounds (wounds that require a daily dressing change)
* osteomyelitis
* systemic infections
* acute Charcot foot and severe chronic Charcot deformity
* ABPI < 0.7 or ankle systolic pressure < 70 mm Hg
* one of the following findings (only 1 out of 3 tests is required):

  * on Doppler waveform analysis on the dorsalis pedis and posterior tibial arteries a monophasic or biphasic flow (with loss of reverse flow) in either foot artery, or
  * a toe: brachial index < 0.7, or
  * transcutaneous oxygen pressure (TcpO2) < 40 mm Hg
* suspicion, presence or history of systemic or local cancer or tumor of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2009-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in ulcer surface area | 4 weeks after treatment start

SECONDARY OUTCOMES:
Incidence of complete wound closure (full re-epithelialization with confirmation 4 weeks afterwards) | At 12 and 16 weeks after treatment start
Incidence of complete wound closure (full re-epithelialization with confirmation 4 weeks afterwards) | Within the whole study period (28 weeks after treatment start)
Time to complete wound closure (full re-epithelialization with confirmation 4 weeks afterwards). | At any time during the study
Incidence of treatment failure defined as <30% decrease in ulcer size | After 8 weeks of treatment
Incidence of patients with ulcer recurrence | Up to 16 and 28 weeks after treatment start
Incidence of treatment-related adverse events (systemic and at the target ulcer) and all AEs/SAEs | During the whole study period
Changes in systemic PDGF-AB and antibody levels against TG-PDGF.AB and aprotinin | At 1, 4, 12, 16 and 20 weeks after treatment start
Changes in vital signs, body weight, physical examination and laboratory parameters | Throughout the study and 28 weeks after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Jamieson, MD, Study Director — Kuros Biosurgery
Locations (34):
- Czechia (4):
  - Diabetologické centrum, I. Interní klinika FN Hradec Králové, Fakultní nemocnice Hradec Králové (21), Hradec Králové
  - Interní klinika 2. Lékařské fakulty UK a FN Motol, Fakultní nemocnice Motol (22), Prague
  - Oddelení diabetologie - Podiatricka ambulance Krajská zdravotní a.s.- Masarykova nemocnice v Ústí nad Labem o.z. (23), Ústí nad Labem
  - Lékařský dum Ormiga Angiologická a diabetologická ambulance (20), Zlín
- Germany (4):
  - Klinikum Sindelfingen-Böblingen (01), Böblingen
  - SRH Klinikum Karlsbad-Langensteinbach (04), Karlsbad
  - Klinikum Stuttgart Bürgerhospital (03), Stuttgart
  - Universitätsklinik Tübingen Chirugische Poliklinik (02), Tübingen
- Hungary (9):
  - Budai Irgalmasrendi Közhasznú Non-Profit Kft (35), Budapest
  - Fõvárosi Önkormányzat Egyesített Szent István és Szent László Kórház - Rendelõintézet Sebészeti Osztály (32), Budapest
  - Fővárosi Önkormányzat Szent Imre Kórház Operativ Szakmák Mátrix Szervezete Általános Sebészeti Profil (33), Budapest
  - Esztergom Város Önkormányzat Vaszary Kolos Kórház Sebészeti Osztály (34), Esztergom
  - Kaposi Mór Oktató Kórház (38), Kaposvár
  - Bács-Kiskun Megyei Önkormányzat Kórháza Szegedi Tudományegyetem Általános Orvostudományi Kar Oktató Kórháza, 2. Belgyógyászat (31), Kecskemét
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház Érsebészeti Osztály (30), Miskolc
  - PTE Klinikai Központ Érsebészeti Klinikai Tanszék (36), Pécs
  - SZTE Szent-Györgyi Albert Klinikai Centrum (37), Szeged
- Romania (5):
  - Institutul Naţional de Diabet, Nutriţie şi Boli Metabolice "Prof. Dr. N. C. Paulescu" (42), Bucharest
  - Spitalul Clinic Judeţean de Urgenţă Cluj (43), Cluj-Napoca
  - Spitalul Clinic Judeţean Mureş, Clinica de Dermatologie (40), Tg Mures
  - Cabinet Medical Individual DermaMed (41), Tg. Mures,
  - Spitalul Clinic Judetean de Urgenta Timisoara (45), Timișoara
- Russia (7):
  - Moscow City Clinical Hospital # 13 (11), Moscow
  - Moscow State University of Public Health "City Clinical (17), Moscow
  - Department of Endocrinology and Diabetes, Russian State Medical University, Moscow City Clinical Hospital # 1 (15), Moscow
  - Department of Diabetic Foot Endocrinology dispensary (12), Moscow
  - Endocrinology Clinic of the State Educational Institute of High Professional Education (18), Moscow
  - Federal State Institution "Federal Bureau of Medical Social Expertise" (10), Moscow
  - Moscow Clinical Hospital # 81 (14), Moscow
- Serbia (5):
  - Klinički centar Srbije, Institut za endokrinologiju, dijabetes i bolesti metabolizma (51), Belgrade
  - Clinical Centre Kragujevac (54), Kragujevac
  - Clinical Centre Nis (50), Niš
  - Clinical Centre of Vojvodina (53), Novi Sad
  - Health Centre Valjevo (52), Valjevo